CLINICAL TRIAL: NCT02506881
Title: International Multicenter Comparative Randomized Double-blind Crossover Study of Pharmacokinetics, Pharmacodynamics and Safety of BCD-066 and Aranesp® After Single Subcutaneous and Intravenous Injection in Healthy Volunteers.
Brief Title: Pharmacokinetics and Pharmacodynamics Study of BCD-066 Compared to Aranesp® in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BCD-066-1
Record Dates: First submitted 2015-07-22; First posted 2015-07-23 (Estimated); Results first posted 2016-05-02 (Estimated); Last update posted 2016-06-14 (Estimated); Status verified 2016-05

CONDITIONS: Healthy
Keywords: darbepoetin alfa; pharmacokinetics; pharmacodynamics; healthy volunteers
MeSH Terms: interventions — Darbepoetin alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- BCD-066 → Aranesp - subcutaneous (Experimental): Volunteers in this group initially will receive a single sc injection of the study drug BCD-066 (darbepoetin alfa) at a dose of 1 µg/kg (on Day 1) and then, after at least 25 days, a single sc injection of the reference drug Aranesp® (darbepoetin alfa) at a dose of 1 µg/kg.
  Interventions: Drug: Darbepoetin alfa
- Aranesp → BCD-066 - subcutaneous (Experimental): Volunteers in this group initially will receive a single sc injection of the reference drug Aranesp® (darbepoetin alfa) at a dose of 1 µg/kg (on Day 1) and then, after at least 25 days, a single sc injection of the study drug BCD-066 (darbepoetin alfa) at a dose of 1 µg/kg.
  Interventions: Drug: Darbepoetin alfa
- BCD-066 → Aranesp - intravenous (Experimental): Volunteers in this group initially will receive a single iv injection of the study drug BCD-066 (darbepoetin alfa) at a dose of 1 µg/kg (on Day 1) and then, after at least 25 days, a single iv injection of the reference drug Aranesp® (darbepoetin alfa) at a dose of 1 µg/kg.
  Interventions: Drug: Darbepoetin alfa
- Aranesp → BCD-066 - intravenous (Experimental): Volunteers in this group initially will receive a single iv injection of the reference drug Aranesp® (darbepoetin alfa) at a dose of 1 µg/kg (on Day 1) and then, after at least 25 days, a single iv injection of the study drug BCD-066 (darbepoetin alfa) at a dose of 1 µg/kg.
  Interventions: Drug: Darbepoetin alfa

INTERVENTIONS:
Drug: Darbepoetin alfa
  Other Names: Aranesp; BCD-066

SUMMARY:
This is a randomized double-blind crossover study of pharmacokinetics, pharmacodynamics and safety of BCD-066 (darbepoetin alfa manufactured by CJSC BIOCAD, Russia) and Aranesp® (Amgen Europe B.V., Netherlands) in healthy volunteers. The purpose of the study is to demonstrate the equivalence of pharmacokinetics, pharmacodynamics and safety parameters after single subcutaneous or intravenous injection. Each drug will be administered to each volunteer at a dose of 1 µg per kilogram as a single subcutaneous or intravenous injection with an interval of at least 25 days.

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* Male gender
* Age 18 - 45 years inclusively
* Body mass index (BMI) 19 - 29 kg/m2 inclusively
* Hemoglobin level 120-160 g/l (12 - 16 g/dL) inclusively during 14 days prior to first study drugs administration
* White blood cells count ≥3,0×109/L, Platelet count ≥140×109/L during 14 days prior to first study drugs administration
* Subjects must be in good health as determined by a medical history, medical examination, electrocardiogram, serum biochemistry, haematology, serology and urinalysis
* Absence of history of systematic alcohol and drug abuse
* Ability of the volunteer, in investigator's opinion, to follow the study protocol procedures and requirements
* Willingness of volunteers and their sexual partners of childbearing potential to use reliable contraception methods starting from 2 weeks before inclusion into the study and until 4 weeks after receiving the last dose of the investigational products. This criterion is not applicable to patients who underwent surgical sterilization. Reliable contraceptive measures include one barrier method in combination with one of the following methods: spermicides, intrauterine device or oral contraceptives used by participant's partner
* Consent to avoid alcohol intake within 24 hours before and 48 hours after each administration of the test or reference drugs

Exclusion Criteria:

* Clinically significant abnormalities on ECG or in laboratory tests, which could interfere with the objective of the study or the safety of the volunteer.
* Clinically significant illness within 4 weeks prior to the screening visit
* Subjects with past or present history of liver disease, angina, renal disease, hypertension, epilepsy, cardiovascular, cerebrovascular, peripheral vascular disease or thrombocytosis
* History of any oncological disease
* Prior exposure to any erythropoietins, darbepoetin
* Prior exposure to IV iron supplementation (within 2 years before randomisation)
* Subjects who have used any medication, including over-the-counter drugs, herbal medications, and nutritional supplements within 14 days prior to IDs administration with the exception of paracetamol (acetaminophen) up to 3g per day or ibuprofen up to 1g per day
* Subjects who smoke more than 10 cigarettes per day
* Subjects who have donated more than 450 ml of blood within the 1 month prior to ID injection
* Epileptic seizures within the 6 months prior to ID injection
* Major surgery within 1 month prior to the enrollment into the study
* Inability to install intravenous catheter (e.g., due to skin disease)
* Subjects who have received any experimental drug within 3 months preceding the 1st ID administration
* Subjects who have a clinically significant history of drug hypersensitivity or allergic disease
* Possibility that the subject will not cooperate with the requirements of the protocol as set out in the volunteer information
* Subjects who consume excessive amounts of caffeine (more than 5 cups of coffee per day)
* Participation in any other clinical study or any preceding participation in other studies within 3 months prior to the 1st ID administration

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Actual)
Dates: Start 2013-03; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Sardaryan, PhD, Principal Investigator — City Mariin Hospital
Locations (1):
- City Mariin Hospital, Saint Petersburg, Russia

RESULTS

PARTICIPANT FLOW:
Groups:
- BCD-066 → Aranesp - Subcutaneous: Volunteers in this group initially will receive a single sc injection of the study drug BCD-066 (darbepoetin alfa) at a dose of 1 µg/kg (on Day 1) and then, after at least 25 days, a single sc injection of the reference drug Aranesp® (darbepoetin alfa) at a dose of 1 µg/kg.
  Darbepoetin alfa
- Aranesp → BCD-066 - Subcutaneous: Volunteers in this group initially will receive a single sc injection of the reference drug Aranesp® (darbepoetin alfa) at a dose of 1 µg/kg (on Day 1) and then, after at least 25 days, a single sc injection of the study drug BCD-066 (darbepoetin alfa) at a dose of 1 µg/kg.
  Darbepoetin alfa
- BCD-066 → Aranesp - Intravenous: Volunteers in this group initially will receive a single iv injection of the study drug BCD-066 (darbepoetin alfa) at a dose of 1 µg/kg (on Day 1) and then, after at least 25 days, a single iv injection of the reference drug Aranesp® (darbepoetin alfa) at a dose of 1 µg/kg.
  Darbepoetin alfa
- Aranesp → BCD-066 - Intravenous: Volunteers in this group initially will receive a single iv injection of the reference drug Aranesp® (darbepoetin alfa) at a dose of 1 µg/kg (on Day 1) and then, after at least 25 days, a single iv injection of the study drug BCD-066 (darbepoetin alfa) at a dose of 1 µg/kg.
  Darbepoetin alfa
Period: First Intervention (Day 1)
Arm/Group | BCD-066 → Aranesp - Subcutaneous | Aranesp → BCD-066 - Subcutaneous | BCD-066 → Aranesp - Intravenous | Aranesp → BCD-066 - Intravenous
Started | 13 | 12 | 25 | 24
Completed | 12 | 12 | 12 | 12
Not Completed | 1 | 0 | 13 | 12
Not completed — Protocol Violation | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0
Not completed — Violation of blood storage conditions | 0 | 0 | 12 | 12
Period: Washout (at Least 25 Days)
Arm/Group | BCD-066 → Aranesp - Subcutaneous | Aranesp → BCD-066 - Subcutaneous | BCD-066 → Aranesp - Intravenous | Aranesp → BCD-066 - Intravenous
Started | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0
Period: Second Intervention (Day 1)
Arm/Group | BCD-066 → Aranesp - Subcutaneous | Aranesp → BCD-066 - Subcutaneous | BCD-066 → Aranesp - Intravenous | Aranesp → BCD-066 - Intravenous
Started | 12 | 12 | 12 | 12
Completed | 12 | 12 | 12 | 12
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Population for safety analysis: all patients who received at least one study drug injection
Groups:
- Total: Total of all reporting groups
Arm/Group | BCD-066 → Aranesp - Subcutaneous | Aranesp → BCD-066 - Subcutaneous | BCD-066 → Aranesp - Intravenous | Aranesp → BCD-066 - Intravenous | Total
Number analyzed (Participants) | 13 | 12 | 25 | 24 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 13 | 12 | 25 | 24 | 74
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 23 [21 to 32] | 22 [21 to 26] | 24 [22 to 27] | 24.5 [21 to 28] | 24 [21 to 28]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0
  Male | 13 | 12 | 25 | 24 | 74

OUTCOME MEASURES:

1. Primary Outcome: AUC
Description: Area Under Concentration-time Curve (AUC) of Darbepoetin Alfa From the Moment of Drug Administration Until 336 (sc administration) or 72 (iv administration) Hours and to Infinity(AUC(0-336)/AUC(0-72) and AUC(0-∞) Respectively Blood samples were taken 30, 20, 10, 0 minutes before injection of study drug and then after 12, 24, 36, 72, 96, 144, 336 and 504 hours post-dose.
Time Frame: 336 hours (sc) / 72 hours (iv)
Population: Population for pharmacokinetics analysis: patients who received at least one study drug injection.
Measure: Median (Inter-Quartile Range); unit: (pg/ml)*hour
Groups:
- BCD-066 Subcutaneous: Pharmacokinetics of darbepoetin alfa after subcutaneous injection of BCD-066 in a dose of 1 µg/kg was analysed.
  AUC of darbepoetin alfa 0 to 336 hours is reported.
- Aranesp® Subcutaneous: Pharmacokinetics of darbepoetin alfa after subcutaneous injection of Aranesp® in a dose of 1 µg/kg was analysed.
  AUC of darbepoetin alfa 0 to 336 hours is reported.
- BCD-066 - Intravenous: Pharmacokinetics of darbepoetin alfa after intravenous injection of BCD-066 in a dose of 1 µg/kg was analysed.
  AUC of darbepoetin alfa 0 to 72 hours is reported.
- Aranesp® - Intravenous: Pharmacokinetics of darbepoetin alfa after intravenous injection of Aranesp® in a dose of 1 µg/kg was analysed.
  AUC of darbepoetin alfa 0 to 72 hours is reported.
Arm/Group | BCD-066 Subcutaneous | Aranesp® Subcutaneous | BCD-066 - Intravenous | Aranesp® - Intravenous
Number analyzed (Participants) | 24 | 24 | 23 | 23
(pg/ml)*hour | 150607 [115435 to 185031] | 152208 [116362 to 212041] | 504584 [463396 to 626538] | 544818 [456106 to 606407]

2. Primary Outcome: Cmax
Description: Maximal concentration of darbepoetin alfa From the Moment of Drug Administration Until 336 (sc administration) or 72 (iv administration) hours.
  Blood samples were taken 30, 20, 10, 0 minutes before injection of study drug and then after 12, 24, 36, 72, 96, 144, 336 and 504 hours post-dose.
Time Frame: 336 hours (sc) / 72 hours (iv)
Population: Population for pharmacokinetics analysis included patients who received at least one study drug injection.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Groups:
- BCD-066 Subcutaneous: Pharmacokinetics of darbepoetin alfa after subcutaneous injection of BCD-066 in a dose of 1 µg/kg was analysed.
  Cmax of darbepoetin alfa 0 to 336 hours is reported.
- Aranesp® Subcutaneous: Pharmacokinetics of darbepoetin alfa after subcutaneous injection of Aranesp® in a dose of 1 µg/kg was analysed.
  Cmax of darbepoetin alfa 0 to 336 hours is reported.
- BCD-066 - Intravenous: Pharmacokinetics of darbepoetin alfa after intravenous injection of BCD-066 in a dose of 1 µg/kg was analysed.
  Cmax of darbepoetin alfa 0 to 72 hours is reported.
- Aranesp® - Intravenous: Pharmacokinetics of darbepoetin alfa after intravenous injection of Aranesp® in a dose of 1 µg/kg was analysed.
  Cmax of darbepoetin alfa 0 to 72 hours is reported.
Arm/Group | BCD-066 Subcutaneous | Aranesp® Subcutaneous | BCD-066 - Intravenous | Aranesp® - Intravenous
Number analyzed (Participants) | 24 | 24 | 23 | 23
pg/ml | 984 [789 to 1226] | 885 [808 to 1197] | 23908 [21535 to 27531] | 24478 [22271 to 29381]

3. Primary Outcome: AUEC
Description: Area Under Effect Curve (AUEC) of reticulocytes count from the Moment of Drug Administration Until 504 hours.
  Blood samples were taken 30, 20, 10, 0 minutes before injection of study drug and then after 12, 24, 36, 72, 96, 144, 336 and 504 hours post-dose.
Time Frame: 504 hours
Population: Population for pharmacokinetics analysis included patients who received at least one study drug injection.
Measure: Median (Inter-Quartile Range); unit: (reticulocytes * 10^9/l)*hour
Groups:
- BCD-066 Subcutaneous: Pharmacodynamics of darbepoetin alfa after subcutaneous injection of BCD-066 in a dose of 1 µg/kg was analysed.
- Aranesp® Subcutaneous: Pharmacodynamics of darbepoetin alfa after subcutaneous injection of Aranesp® in a dose of 1 µg/kg was analysed.
- BCD-066 - Intravenous: Pharmacodynamics of darbepoetin alfa after intravenous injection of BCD-066 in a dose of 1 µg/kg was analysed.
- Aranesp® - Intravenous: Pharmacodynamics of darbepoetin alfa after intravenous injection of Aranesp® in a dose of 1 µg/kg was analysed.
Arm/Group | BCD-066 Subcutaneous | Aranesp® Subcutaneous | BCD-066 - Intravenous | Aranesp® - Intravenous
Number analyzed (Participants) | 24 | 24 | 23 | 23
(reticulocytes * 10^9/l)*hour | 28248 [22162 to 32648] | 27916 [22827 to 32628] | 35610 [29578 to 41423] | 36928 [28773 to 42247]

4. Primary Outcome: AC-Emax
Description: Maximum elevation of absolute reticulocyte count from the baseline from the Moment of Drug Administration Until 504 hours.
  Blood samples were taken 30, 20, 10, 0 minutes before injection of study drug and then after 12, 24, 36, 72, 96, 144, 336 and 504 hours post-dose.
Time Frame: 504 hours
Population: Population for analysis of pharmacodynamics included patients who received at least one study drug injection.
Measure: Median (Inter-Quartile Range); unit: reticulocytes * 10^9/l
Arm/Group | BCD-066 Subcutaneous | Aranesp® Subcutaneous | BCD-066 - Intravenous | Aranesp® - Intravenous
Number analyzed (Participants) | 24 | 24 | 23 | 23
reticulocytes * 10^9/l | 44.8 [26.8 to 62.3] | 54.55 [40.7 to 69.0] | 71.3 [51.9 to 85.3] | 72.1 [55.5 to 86.7]

5. Secondary Outcome: T1/2
Description: Serum half-life of darbepoetin alfa after single sc of iv administration. Blood samples were taken 30, 20, 10, 0 minutes before injection of study drug and then after 12, 24, 36, 72, 96, 144, 336 and 504 hours post-dose.
Time Frame: 336 hours (sc) / 72 hours (iv)
Population: Population for pharmacokinetics analysis: patients who received at least one study drug injection.
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | BCD-066 Subcutaneous | Aranesp® Subcutaneous | BCD-066 - Intravenous | Aranesp® - Intravenous
Number analyzed (Participants) | 24 | 24 | 23 | 23
hours | 74.8 [69.6 to 92.6] | 80.6 [65.7 to 89.9] | 13.1 [12.7 to 13.9] | 12.7 [12.4 to 13.9]

6. Secondary Outcome: Tmax
Description: Time to achieve maximum serum concentration of darbepoetin alfa after single sc of iv administration
Time Frame: 336 hours (sc) / 72 hours (iv)
Population: Population for pharmacokinetics analysis: patients who received at least one study drug injection.
Measure: Median (Inter-Quartile Range); unit: hours
Groups:
- BCD-066 - Subcutaneous: Pharmacodynamics of darbepoetin alfa after subcutaneous injection of BCD-066 in a dose of 1 µg/kg was analysed.
- Aranesp® - Subcutaneous: Pharmacodynamics of darbepoetin alfa after subcutaneous injection of Aranesp® in a dose of 1 µg/kg was analysed.
Arm/Group | BCD-066 - Subcutaneous | Aranesp® - Subcutaneous | BCD-066 - Intravenous | Aranesp® - Intravenous
Number analyzed (Participants) | 24 | 24 | 23 | 23
hours | 36 [16 to 36] | 36 [36 to 36] | 0.25 [0.08 to 0.50] | 0.25 [0.08 to 0.40]

7. Secondary Outcome: Cl
Description: Serum clearance of of darbepoetin alfa after single sc of iv administration. Blood samples were taken 30, 20, 10, 0 minutes before injection of study drug and then after 12, 24, 36, 72, 96, 144, 336 and 504 hours post-dose.
Time Frame: 336 hours (sc) / 72 hours (iv)
Population: Population for pharmacokinetics analysis: patients who received at least one study drug injection.
Measure: Median (Inter-Quartile Range); unit: hours*kg
Arm/Group | BCD-066 - Subcutaneous | Aranesp® - Subcutaneous | BCD-066 - Intravenous | Aranesp® - Intravenous
Number analyzed (Participants) | 24 | 24 | 23 | 23
hours*kg | 0.433 [0.308 to 0.587] | 0.375 [0.314 to 0.566] | 139.0 [123.9 to 153.7] | 134.2 [114.0 to 159.2]

ADVERSE EVENTS:
Time Frame: 0 to 504 hours after injection
Groups:
- BCD-066 Subcutaneous: Safety parameters of darbepoetin alfa after subcutaneous injection of BCD-066 in a dose of 1 µg/kg are presented.
- Aranesp® Subcutaneous: Safety parameters of darbepoetin alfa after subcutaneous injection of Aranesp® in a dose of 1 µg/kg are presented.
- BCD-066 - Intravenous: Safety parameters of darbepoetin alfa after intravenous injection of BCD-066 in a dose of 1 µg/kg are presented.
- Aranesp® - Intravenous: Safety parameters of darbepoetin alfa after intravenous injection of Aranesp® in a dose of 1 µg/kg are presented.
Arm/Group | BCD-066 Subcutaneous | Aranesp® Subcutaneous | BCD-066 - Intravenous | Aranesp® - Intravenous
Serious Adverse Events (participants affected / at risk) | 0/25 | 0/25 | 0/49 | 0/49
Other Adverse Events (participants affected / at risk) | 23/25 | 22/25 | 44/49 | 42/49
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BCD-066 Subcutaneous (N=25) | Aranesp® Subcutaneous (N=25) | BCD-066 - Intravenous (N=49) | Aranesp® - Intravenous (N=49)
Anemia (Blood and lymphatic system disorders) | 2 | 1 | 2 | 2
Elevated hematocrit (Blood and lymphatic system disorders) | 1 | 2 | 3 | 4
Elevated reticulocyte count (Blood and lymphatic system disorders) | 17 | 17 | 41 | 42
Leucopenia (Blood and lymphatic system disorders) | 5 | 5 | 5 | 5
Leucocytosis (Blood and lymphatic system disorders) | 9 | 6 | 11 | 17
Neutropenia (Blood and lymphatic system disorders) | 5 | 6 | 7 | 6
Decrease in hematocrit (Blood and lymphatic system disorders) | 2 | 2 | 6 | 5
Decrease in reticulocyte count (Blood and lymphatic system disorders) | 6 | 7 | 9 | 4
Trombocytopenia (Blood and lymphatic system disorders) | 4 | 3 | 6 | 9
Monocytosis (Blood and lymphatic system disorders) | 10 | 11 | 28 | 19
Elevated neutrophil count (Blood and lymphatic system disorders) | 2 | 1 | 5 | 6
Elevated basophil count (Blood and lymphatic system disorders) | 2 | 1 | 1 | 2
Decreased eosinophil count (Blood and lymphatic system disorders) | 1 | 2 | 0 | 1
Increased eosinophil count (Blood and lymphatic system disorders) | 2 | 1 | 4 | 6
Elevated creatinine (Renal and urinary disorders) | 2 | 1 | 5 | 7
Erythrocytosis (Blood and lymphatic system disorders) | 1 | 0 | 12 | 13
Trombocytosis (Blood and lymphatic system disorders) | 0 | 1 | 4 | 5
Elevated ALT (Hepatobiliary disorders) | 1 | 1 | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No